CLINICAL TRIAL: NCT01101490
Title: Changes of Right and Left Cerebral Oxygen Saturation and Blood Flow During Nephrectomy in Lateral Decubitus Position
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Jeong-Yeon Hong / instructor, Yonsei University, College of Medicine
Other Study IDs: 4-2009-0724
Record Dates: First submitted 2010-04-08; First posted 2010-04-12 (Estimated); Last update posted 2011-04-22 (Estimated); Status verified 2011-04

CONDITIONS: Nephrectomy
Keywords: To compare the change of cerebral oxygen saturation and blood flow between right and left side in lateral decubitus position during nephrectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine changes of right and left cerebral oxygen saturation and blood flow during nephrectomy in lateral decubitus position.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (ASA physical status I and II) aged between 20-65 yrs

Exclusion Criteria:

* Cardiovascular, renal, hepatic disease, or communication failure

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the patients who visit Severance hospital for nephrectomy
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-04; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
brain oximeter saturation(%) | 1 hour after operation
blood flow | 1 hour after operation
velocity of superficial temporal artery in right and left side | 1 hour after operation

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-Yeon Hong, Principal Investigator — Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, Korea
Locations (1):
- Severance Hospital, Department of Anesthesiology & Pain Medicine, Seoul, South Korea